CLINICAL TRIAL: NCT03185676
Title: The Long Term Efficacy of a Bilberry-based Probiotic Product on Glucose Tolerance and Insulin Resistance as Compared to a Control.
Brief Title: Efficacy of a Bilberry-based Probiotic Product on Glucose Tolerance and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Åsa Håkansson, Associate Senior Lecturer, Lund University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: InVeg (2)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Vaccinium myrtillus extract; Beverages; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Billberry (Experimental): A bilberry-based probiotic beverage
  Interventions: Other: Bilberry
- Control (Active Comparator): A control beverage without bilberries or probiotics
  Interventions: Other: beverage without bilberries or probiotics

INTERVENTIONS:
Other: Bilberry — A bilberry based probiotic beverage
  Arms: Billberry
Other: beverage without bilberries or probiotics — A control beverage without bilberries or probiotics
  Arms: Control

SUMMARY:
The impact of a bilberry-based probiotic drink on the postprandial levels of serum glucose and insulin have already been study in the past. The aim of the current study is to evaluate the long term effect of the probiotic bilberry drink on glucose tolerance and insulin resistance in healthy adults and in comparison to a control drink.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults with a BMI between 20-30

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
The long term effect of a bilberry-based probiotic beverage on postprandial levels of serum insulin | Incremental area under the curve for serum insulin from 0 min up to 120 min following the ingestion of the study product
  The incremental area under the curve (AUC) will be measured for the levels of postprandial serum insuling from 0 min to 120 min following ingestion of the product (included intermediate measuring time points are 30, 60 and 90 min)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinisk Prövningsenhet, Kliniska Studier Sverige - Forum Söder, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No